CLINICAL TRIAL: NCT00329082
Title: LY2062430: Multiple-Dose Safety in Subjects With Mild-to-Moderate Alzheimer's Disease and Single-Dose Safety in Healthy Volunteers
Brief Title: Effects of LY2062430 in Subjects With Mild-to-Moderate Alzheimer's Disease and in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6649; H8A-MC-LZAJ
Record Dates: First submitted 2006-05-19; First posted 2006-05-24 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — solanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: LY2062430
- 2 (Experimental)
  Interventions: Drug: LY2062430
- 3 (Experimental)
  Interventions: Drug: LY2062430
- 4 (Experimental)
  Interventions: Drug: LY2062430
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2062430 — 1. 100mg QW IV for 12 weeks
  2. 100mg Q4W IV for 12 weeks
  3. 400mg QW IV for 12 weeks
  4. 400mg Q4W IV for 12 weeks
  Arms: 1; 2; 3; 4
Drug: Placebo — 5: Placebo QW IV for 12 weeks
  Arms: 5

SUMMARY:
To study the safety of LY2062430 in patients with mild-to-moderate Alzheimer's disease and in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* At least 50 years of age and diagnosed with mild to moderate Alzheimer's disease or healthy volunteers
* fluent in reading and speaking English
* AD patients must have a reliable study partner who will be in frequent contact with the patient and comply with protocol requirements
* AD patients who have received AChEIs or memantine for at least 4 months and on stable therapy for at least 2 months prior to starting study drug

Exclusion Criteria:

* Have a history of serious infectious disease affecting the brain, head trauma, cancer, drug or alcohol abuse in the past 5 years
* Have serious or uncontrolled health problems or laboratory tests
* Multiple or severe drug allergies
* Prior participation in an active immunization study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 1 year

SECONDARY OUTCOMES:
To determine the plasma pharmacokinetics of LY2062430 | 1 year
To evaluate the pharmacokinetic/pharmacodynamic relationships between LY2062430 concentrations and plasma peptide amyloid beta concentrations | 1 year
To evaluate the changes in thinking and memory | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com